CLINICAL TRIAL: NCT03478358
Title: Treatment of a Long-lasting Radiolabeled Somatostatin Analogue 177Lu-DOTA-EB-TATE in Patients With Advanced Metastatic Neuroendocrine Tumors
Brief Title: Treatment Using 177Lu-DOTA-EB-TATE in Patients With Advanced Neuroendocrine Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-NM018
Record Dates: First submitted 2018-02-05; First posted 2018-03-27 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — (177)Lu-DOTA-EB-TATE; Amino Acids; Lysine; Arginine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 177Lu-DOTA-EB-TATE 1 (Experimental): The patients were intravenously injected with single dose 0.37GBq-0.74GBq (10-30 mCi) of 177LuDOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-DOTA-EB-TATE 1
- 177Lu-DOTA-EB-TATE 2 (Experimental): The patients were intravenously injected with single dose 1.85GBq (50 mCi) of 177LuDOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-DOTA-EB-TATE 2
- 177Lu-DOTA-EB-TATE 3 (Experimental): The patients were intravenously injected with single dose 3.7 GBq (100 mCi) of 177LuDOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-DOTA-EB-TATE 3
- 177Lu-DOTA-TATE (Experimental): The patients were intravenously injected with single dose 3.7 GBq (100 mCi) of 177LuDOTA-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-DOTA-TATE
- 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE with amino acids (lysine and arginine) (Experimental): The patients were intravenously injected with 3.7 GBq (100 mCi) of 177LuDOTA-TATE and amino acids (lysine and arginine).
  Interventions: Drug: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE with amino acids (lysine and arginine)
- 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE without amino acids (lysine and arginine) (Experimental): The patients were intravenously injected with 3.7 GBq (100 mCi) of 177LuDOTA-TATE without amino acids (lysine and arginine).
  Interventions: Drug: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE without amino acids (lysine and arginine)

INTERVENTIONS:
Drug: 177Lu-DOTA-EB-TATE 1 — The patients were intravenously injected with single dose 0.37GBq-0.74GBq (10-30 mCi) of 177Lu-DOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Arms: 177Lu-DOTA-EB-TATE 1
Drug: 177Lu-DOTA-TATE — The patients were intravenously injected with single dose 3.7GBq (100 mCi) of 177Lu-DOTA-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Arms: 177Lu-DOTA-TATE
Drug: 177Lu-DOTA-EB-TATE 2 — The patients were intravenously injected with single dose 1.85GBq (50 mCi) of 177Lu-DOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Arms: 177Lu-DOTA-EB-TATE 2
Drug: 177Lu-DOTA-EB-TATE 3 — The patients were intravenously injected with single dose 3.7GBq (100 mCi) of 177Lu-DOTA-EB-TATE and underwent 68Ga-DOTATATE PET/CT scans before and after the treatment.
  Arms: 177Lu-DOTA-EB-TATE 3
Drug: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE with amino acids (lysine and arginine) — The patients were intravenously injected with 3.7GBq (100 mCi) of 177Lu-DOTA-EB-TATE and amino acids (lysine and arginine).
  Arms: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE with amino acids (lysine and arginine)
Drug: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE without amino acids (lysine and arginine) — The patients were intravenously injected with 3.7GBq (100 mCi) of 177Lu-DOTA-EB-TATE without amino acids (lysine and arginine).
  Arms: 3.7 GBq (100 mCi) of 177Lu-DOTA-EB-TATE without amino acids (lysine and arginine)

SUMMARY:
This is a prospective study to investigate the long-lasting radiolabeled somatostatin analogue based peptide receptor radionuclide therapy and evaluate response to 177Lu-DOTA-EB-TATE in patients with advanced metastatic neuroendocrine tumors. Different groups with doses of 0.37GBq-0.74GBq (10-20 mCi) and 1.85GBq (50 mCi)of 177Lu-DOTA-EB-TATE, 3.7GBq (100 mCi)of 177Lu-DOTA-TATE will be injected intravenously. Besides, we evaluated the safety and dosimetry of 3.7GBq (100 mCi) of 177Lu-DOTA-EB-TATE with and without amino acid infusion. All patients will undergo 68Ga-DOTATATE PET/CT scans before and after the treatment.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a heterogeneous group of neoplasms that can develop anywhere in the body and arise from neuroendocrine cells throughout the endocrine system. The most recent NCCN guidelines for unresectable and metastatic NET recommend somatostatin analogues as first-line treatment, but do not recommend a particular treatment sequence for the remaining therapies. Radiolabeled somatostatin analogue therapy, also known as peptide receptor radionuclide therapy has become a well-accepted treatment for patients with well to moderately differentiated unresectable or metastatic NETs and disease progression after first-line treatment. However, a major problem in the therapeutic use of 177Lu-Dotatate has been its short half-life and fast rate of clearance. Kidney is considered one of the dose-limiting organs in peptide receptor radionuclide therapy (PRRT). Amino acid has been infused to reduce renal absorbed dose by inhibiting the proximal tubular reabsorption of the radiopeptide. This study was designed to compare the efficacy of a long-lasting radiolabeled somatostatin analogue 177Lu-DOTA-EB-TATE with 177Lu-DOTA-TATE in patients with advanced metastatic neuroendocrine tumors and evaluate the safety and dosimetry of 3.7GBq (100 mCi) of 177Lu-DOTA-EB-TATE with and without amino acid infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adults who had neuroendocrine tumors and had metastasized, that were with histologically confirmed, inoperable and had showed disease progression according to Response Evaluation Criteria in Solid Tumors [RECIST]. Tumors were with well-differentiated histologic features and a Ki67 index of 0 to 20%. Target tumors were selected from CT, MRI, and 68Ga-DOTA-TATE PET/CT, with confirmed somatostatin receptorexpressing and at least one lesion has higher uptake than that of normal liver parenchyma on 68Ga-DOTA-TATE PET imaging within 1 weeks.

Exclusion Criteria:

* The exclusion criteria were a serum creatinine level of more than 150 μmol per liter, baseline measured GFR of less than 50 mL/min/1.73 m2, determined by 99mTc-DTPA renal function examination, a hemoglobin level of less than 8.0 g/dl, a white-cell count of less than 2.0× 109/L, a platelet count of less than 75 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia, and pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of standardized uptake value of 68Ga-DOTA-TATE before and after the treatment in metastatic neuroendocrine tumors | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value before and after the treatment in metastatic neuroendocrine tumors will be measured.
the safety of 3.7GBq of 177Lu-DOTA-EB-TATE with and without amino acid infusion. | 1 year
  Hematological parameters, liver, and renal function at baseline, 1 week and 4 weeks after PRRT were tested. 99mTc-DTPA dynamic renal imaging for the determination of the glomerular filtration rate (GFR) was performed at baseline and 8 weeks after each cycle of PRRT.

SECONDARY OUTCOMES:
the dosimetry of 3.7GBq of 177Lu-DOTA-EB-TATE with and without amino acid infusion. | 1 year
  the absorbed dose for kidney and whole-body evaluated through HERMES software.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, M.D.,PhD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Jiang Y, Liu Q, Wang G, Zhang J, Zhu Z, Chen X. Evaluation of Safety, Biodistribution, and Dosimetry of a Long-Acting Radiolabeled Somatostatin Analog 177 Lu-DOTA-EB-TATE With and Without Amino Acid Infusion. Clin Nucl Med. 2023 Jun 1;48(6):e289-e293. doi: 10.1097/RLU.0000000000004642. Epub 2023 Apr 18. PMID 37075254
- [Derived] Liu Q, Cheng Y, Zang J, Sui H, Wang H, Jacobson O, Zhu Z, Chen X. Dose escalation of an Evans blue-modified radiolabeled somatostatin analog 177Lu-DOTA-EB-TATE in the treatment of metastatic neuroendocrine tumors. Eur J Nucl Med Mol Imaging. 2020 Apr;47(4):947-957. doi: 10.1007/s00259-019-04530-1. Epub 2019 Dec 12. PMID 31832728